CLINICAL TRIAL: NCT01397097
Title: Multicenter, Open-label, Randomized, Controlled Parallel-group Study to Assess Discontinuation Rates, Bleeding Patterns, User Satisfaction and Adverse Event Profile of LCS12 in Comparison to Etonorgestrel Subdermal Implant Over 12 Months of Use in Women 18 to 35 Years of Age
Brief Title: LCS12 vs. ENG Subdermal Implant (Nexplanon) Discontinuation Rate Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13363; 2010-023911-32 (EudraCT Number)
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Contraception
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: LNG-IUS (BAY 86-5028)
- Arm 2 (Active Comparator)
  Interventions: Drug: 68 mg etonorgestrel implant for subdermal use (Nexplanon)

INTERVENTIONS:
Drug: LNG-IUS (BAY 86-5028) — LCS12 insertion will occur at randomization visit (Visit 2). Duration of study treatment is 12 months with an follow-up extension for up to 3 years
  Arms: Arm 1
Drug: 68 mg etonorgestrel implant for subdermal use (Nexplanon) — Implant insertion will occur at randomization visit (Visit 2). Duration of study treatment is 12 months, may be continued up to 3 years under standard care.
  Arms: Arm 2

SUMMARY:
The primary objective is to demonstrate that discontinuation rates in women (ages 18-35 years inclusive) using LCS12 are not higher than those seen in women using ENG subdermal implant over a period of 12 months.

Secondary objectives are to observe the bleeding patterns, adverse event profiles and the occurrence of unintended pregnancies. Additionally, data on user satisfaction, IUS expulsions and implant site complications will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated the informed consent
* Healthy female subjects in need of contraception
* Age: between 18 and 35 years (inclusive) at Screening visit
* Normal or clinically insignificant cervical smear not requiring further follow up (a cervical smear has to be taken at screening visit or a normal result has to be documented within the previous six months). HPV testing in subjects with ASCUS can be used as an adjunctive test. Subjects with ASCUS can be included if they are negative for high-risk HPV strains.
* History of regular cyclic menstrual periods as determined by subject's history, subject has regular menstrual cycles (length of cycle 21 - 35 days). (Subject's history while not using hormonal contraceptives is sufficient, no washout period is required).
* Subject is willing and able to attend the scheduled study visits and to comply with the study procedures.

Exclusion Criteria:

* Pregnancy or currently lactating
* Vaginal delivery, cesarean delivery or abortion within 6 weeks prior to Screening visit. Note: Postpartum LCS12 insertions should be postponed until uterus is fully involuted, however not earlier than 6 weeks after delivery. If involution is substantially delayed, consider waiting until 12 weeks postpartum.
* Infected abortion or postpartum endometritis within 3 months prior to the Screening visit.
* Undiagnosed abnormal genital bleeding.
* Acute lower genital tract infection (until successfully treated)
* Acute or history of recurrent, pelvic inflammatory disease.
* Congenital or acquired uterine anomaly or any distortion of the uterine cavity (e.g. by fibroids) that, in the opinion of the investigator or designee, would cause problems during insertion, retention, or removal of LCS12. (Note: a pre-insertion ultrasound is not necessary. However, if based on subject history or physical exam findings, there is a suspicion of uterine anomaly or any distortion of the uterine cavity, appropriate diagnostic measures should be taken prior to randomization)
* History of, diagnosed or suspected genital malignancy, and untreated cervical dysplasia.
* Clinically significant endometrial polyp(s) that, in the opinion of the investigator or designee, may interfere with the assessment of the bleeding profile during the study. (Note: a pre-insertion ultrasound is not necessary. However, if based on subject history or physical exam findings, there is a suspicion of polyps, appropriate diagnostic measures should be taken prior to randomization.)
* Has previously failed screening for this study
* Any disease or condition that may worsen under hormonal treatment according to the assessment and opinion of the investigator. The following are examples of such conditions or diseases:

  * Cardiovascular
  * Presence or a history of venous or arterial thrombotic/thromboembolic events (e.g., deep venous thrombosis, pulmonary embolism, myocardial infarction) or of a cerebrovascular accident, including prodromi (e.g. transient ischemic attack, angina pectoris)
  * Repeated measurements of systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg.

Liver

* Presence or history of liver tumors (benign or malignant)
* Presence or history of severe hepatic disease as long as liver function values have not returned to normal
* Jaundice and/or pruritus related to cholestasis (Gilbert's syndrome excepted)
* History of cholestatic jaundice associated with pregnancy or previous COC use

  - Other diseases:
* Malignant or premalignant disease (excluding melanoma)
* History of migraine with focal neurologic symptoms

  * Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
  * Clinically significant ovarian cyst (defined as abnormal non-functional cysts) (Note: a pre-insertion ultrasound is not necessary. However, if based on subject history or physical exam findings, there is a suspicion of a clinically significant cyst, appropriate diagnostic measures should be taken prior to randomization.)
  * Any diseases or conditions that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism or altered excretion of the study medication
  * Other contraceptive methods:
* Sterilization
* Use of any long-acting injectable sex-hormone preparations within 10 months prior to the Randomization visit. The use of non study oral, vaginal, or transdermal hormonal contraception, intrauterine devices (IUDs) with or without hormonal release, and implants is prohibited during treatment.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 766 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Discontinuation rate by treatment group | at 12 months

SECONDARY OUTCOMES:
Discontinuation rates by treatment group | at 6 months and by reason at 6 and 12 months
Overall satisfaction rating and questionnaires on User satisfaction and bleeding and Contraceptive tolerability | at 6 and 12 months
Pregnancy rate, as determined by Pearl index | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (37):
- Australia (5):
  - Ashfield, New South Wales
  - Sydney, New South Wales
  - North Adelaide, South Australia
  - Parkville, Victoria
  - Nedlands, Western Australia
- Finland (6):
  - Espoo
  - Helsinki
  - Kuopio
  - Tampere
  - Tampereen Yliopisto
  - Turku
- France (8):
  - Biarritz
  - Bordeaux
  - Marseille
  - Quetigny
  - Reims
  - Schiltigheim
  - Seclin
  - Strasbourg
- Norway (5):
  - Elverum
  - Haugesund
  - Ski
  - Straume
  - Trondheim
- Sweden (7):
  - Gothenburg
  - Linköping
  - Luleå
  - Malmo
  - Örebro
  - Stockholm
  - Uppsala
- United Kingdom (6):
  - Cambridge, Cambridgeshire
  - London, London
  - Sheffield, South Yorkshire
  - Leeds, West Yorkshire
  - Liverpool
  - London

REFERENCES:
- [Derived] Apter D, Briggs P, Tuppurainen M, Grunert J, Lukkari-Lax E, Rybowski S, Gemzell-Danielsson K. A 12-month multicenter, randomized study comparing the levonorgestrel intrauterine system with the etonogestrel subdermal implant. Fertil Steril. 2016 Jul;106(1):151-157.e5. doi: 10.1016/j.fertnstert.2016.02.036. Epub 2016 Mar 24. PMID 27016644